CLINICAL TRIAL: NCT00121719
Title: An Open Label Phase I Dose Escalation Study Of E7080
Brief Title: An Open Label Dose Escalation Study Of E7080
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-E044-101; 2004-002265-21 (EudraCT Number)
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor or Lymphoma
Keywords: Resistant and refractory solid tumors; lymphomas; hodgkins disease; non-hodgkins lymphoma; neoplasms
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms | interventions — lenvatinib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib tablets taken orally, once daily.
  Other Names: E7080

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of lenvatinib in patients with solid tumors or lymphomas.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, dose escalation study. Patients will be treated with lenvatinib once daily. Each four-week treatment period will be considered to be one treatment cycle. The selection of subsequent dose levels will be performed according to an accelerated design: Although initially 3 patients per dose level will be entered, the next dose level can be opened for patient accrual after only the first patient in the previous cohort completes Cycle 1 with no drug-related toxicity greater than grade 1 (except alopecia, lymphopenia and anemia).

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet all of the inclusion criteria outlined below in order to be eligible to participate in the study:

1. Patients with histologically and/or cytologically confirmed solid tumor or lymphoma who are resistant/refractory to approved therapies or for whom no appropriate therapies are available.
2. All previous treatment (including surgery and radiotherapy) must have been completed at least four weeks prior to study entry and any acute toxicities must have resolved.
3. Aged greater than or equal to 18 years.
4. Karnofsky performance status greater than or equal 70%.
5. Written informed consent to participate in the study.

EXCLUSION CRITERIA:

Patients with the following characteristics will not be eligible for the study:

1. Brain tumors or brain or leptomeningeal metastases.
2. Any of the following laboratory parameters:

   1. hemoglobin less than 9 g/dl (5.6 mmol/L)
   2. neutrophils less than 1.5 x 10^9/L
   3. platelets less than 100 x 10^9/L
   4. serum bilirubin greater than 25 micro-mol/l (1.5 mg/dl)
   5. other liver parameters greater than 3 x the upper limit of normal (ULN)
   6. serum creatinine greater than 1.5 x ULN or creatinine clearance less than 60 ml/minute
3. Uncontrolled infections.
4. Clinically significant cardiac impairment or unstable ischemic heart disease including a myocardial infarction within six months of study start.
5. Any treatment with investigational drugs within 30 days before the start of the study.
6. Pregnancy or lactation (all women of childbearing potential must have a negative pregnancy test before inclusion in the study; post-menopausal women must be amenorrheic for at least 12 months). Female patients of childbearing potential must use adequate contraceptive protection, defined as two forms of contraception, one of which must be a barrier method.
7. Fertile males not willing to use contraception or whose female partners are not using adequate contraceptive protection.
8. History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the investigator, would impair study compliance.
9. Legal incapacity.
10. Centrally located or squamous cell carcinoma of the lung.
11. Proteinuria greater than 1+ on bedside testing.
12. History of gastrointestinal malabsorption.
13. Surgery involving gastro- and/or intestinal anastomosis within four weeks of study start.
14. Patients with bleeding or thrombotic disorders.
15. Patients using therapeutic dosages of anticoagulants.
16. Poorly controlled hypertension (defined as a change in hypertensive therapy within three months of study start) or patients diagnosed with hypertension (defined as a repeat blood pressure measurement of 160/90 mmHg or higher) at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-07-01 (Actual); Primary Completion 2009-06-19 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands Cancer Institute- Antoni Van Leeuwenhoek Hospital, Amsterdam, Netherlands
- Gartnavel General Hospital, Glasgow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 site in United Kingdom and 1 site in Netherlands from 01 July 2005 to 01 March 2019.
Pre-assignment Details: A total of 82 participants with solid tumors or lymphomas were enrolled and received study treatment.
Groups:
- Lenvatinib 0.2 mg: Two 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced dose-limiting toxicity (DLT) during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the maximum tolerated dose (MTD) was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 0.4 mg: Four 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 0.8 mg: Eight 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 1.6 mg: One 1.0 mg lenvatinib tablet and six 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 3.2 mg: Three 1.0 mg lenvatinib tablets and two 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 6.4 mg: Six 1.0 mg lenvatinib tablets and four 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 12 mg: One 10 mg lenvatinib tablet and two 1.0 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 12.5 mg: One 10 mg lenvatinib tablet, two 1.0 mg lenvatinib tablets, and five 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 16 mg: One 10 mg lenvatinib tablet and six 1.0 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 20 mg: Two 10 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib Fasted/Fed 25 mg: Participants from the MTD Cohort who chose to participate in the food-effect pilot study were randomly assigned to this Cohort. Two 10 mg lenvatinib tablets and five 1.0 mg lenvatinib tablets were taken orally, once daily. The Day 15 dose of lenvatinib was taken in a fasted state and the Day 22 dose was taken in a fed state with a high fat meal. All other doses were taken on an empty stomach after waking, followed by fasting for 2 hours with only clear liquids allowed.
- Lenvatinib Fed/Fasted 25 mg: Participants from the MTD Cohort who chose to participate in the food-effect pilot study were randomly assigned to this Cohort. Two 10 mg lenvatinib tablets and five 1.0 mg lenvatinib tablets were taken orally, once daily. The Day 15 dose of lenvatinib was taken in a fed state with a high fat meal and the Day 22 dose was taken in a fasted state. All other doses were taken on an empty stomach after waking, followed by fasting for 2 hours with only clear liquids allowed.
- Lenvatinib (MTD Cohort) 25 mg: Participants in this cohort had the option of participating in the food-effect pilot study. Two 10 mg lenvatinib tablets and five 1.0 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
- Lenvatinib 32 mg: Three 10 mg lenvatinib tablets and two 1.0 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
Period: Dose Escalation (4 Weeks)
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib Fasted/Fed 25 mg | Lenvatinib Fed/Fasted 25 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Started | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 0 | 0 | 24 | 7
Completed | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 0 | 0 | 24 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Food-Effect Pilot Study (4 Weeks)
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib Fasted/Fed 25 mg | Lenvatinib Fed/Fasted 25 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of lenvatinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (7.94) | 47.8 (6.45) | 64.0 (6.48) | 60.0 (11.53) | 65.0 (19.00) | 51.0 (22.72) | 46.3 (13.25) | 52.6 (13.28) | 55.7 (13.32) | 51.7 (12.34) | 52.2 (9.65) | 53.9 (11.84) | 53.4 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 1 | 2 | 0 | 8 | 3 | 3 | 0 | 14 | 1 | 39
  Male | 2 | 1 | 2 | 2 | 1 | 3 | 4 | 6 | 3 | 3 | 10 | 6 | 43

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose level at which no more than one out of six participants experienced dose-limiting toxicity (DLT). DLT was assessed during the first 4 weeks of therapy (Cycle 1) for dose escalation purposes. Participants enrolled into the MTD cohort were given the option to also participate in the food-effect pilot study. The food-effect pilot study was initiated once the MTD had been established.
Time Frame: Cycle 1 (4 weeks)
Population: ITT population included all participants who received at least one dose of lenvatinib.
Measure: Number; unit: milligram (mg)
Groups:
- Lenvatinib: Participants not in the food-effect pilot study: 25 mg lenvatinib was administered orally once daily on an empty stomach shortly after waking. Participants fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this period. Grapefruit juice was to be avoided during the study.
  Participants in the food-effect pilot study: 25 mg lenvatinib was administered as described above except on Days 15 and 22 in Cycle 1. Participants in this pilot study were randomly assigned to receive lenvatinib under a fed state (following a high fat meal) or fasting state (overnight fast greater than or equal to 10 hours) on Day 15, then in the reverse/untried state on Day 22. For both cases, no food was allowed for 4 hour following administration of lenvatinib.
Arm/Group | Lenvatinib
Number analyzed (Participants) | 82
milligram (mg) | 25

2. Secondary Outcome: Summary of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: All AEs were graded on a 5-point scale according to the National Cancer Institute's Common Toxicity Criteria (NCI CTC) grading system, version 3.0. Safety was assessed using the occurrence of DLTs, AEs, SAEs, clinical laboratory test results, vital signs measurements, physical examination findings, and electrocardiograms (ECGs) readings. An AE was defined as any untoward medical occurrence in a participant administered lenvatinib and did not necessarily have a causal relationship to lenvatinib. An SAE was defined as any untoward medical occurrence which results in death, was life-threatening, required hospitalization or prolonged hospitalization, resulted in persistent or significant disability/incapacity, or caused a congenital anomaly/birth defect. Treatment-related AEs and SAEs are AEs considered probably or possibly related to lenvatinib.
Time Frame: First date of study treatment to date of last dose of study treatment, up to approximately 13 years and 8 months
Population: Safety population (ITT population) included all participants who received at least one dose of lenvatinib.
Measure: Number; unit: Percentage of participants
Groups:
- Lenvatinib 0.2 mg: Two 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and the MTD was determined. An additional 12 participants were treated at the MTD level.
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib Fasted/Fed 25 mg | Lenvatinib Fed/Fasted 25 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 6 | 5 | 24 | 7
Percentage of participants
  Adverse events | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Treatment-related adverse events | 75.0 | 75.0 | 50.0 | 66.7 | 100.0 | 100.0 | 91.7 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 85.7
  Serious adverse events | 50.0 | 50.0 | 25.0 | 33.3 | 0 | 100.0 | 41.7 | 44.4 | 33.3 | 100.0 | 33.3 | 40.0 | 62.5 | 42.9
  Treatment-related serious adverse events | 25.0 | 0 | 25.0 | 0 | 0 | 33.3 | 8.3 | 11.1 | 33.3 | 66.7 | 16.7 | 20.0 | 33.3 | 14.3

3. Secondary Outcome: Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any grade 3 or higher hematological or non-hematological toxicity directly related to lenvatinib, any repeated National Cancer Institute Common Toxicity Criteria (NCI CTC) grade 2 hematological or non-hematological toxicity considered to be directly related to lenvatinib and required dose reduction, or failure to administer greater than or equal to 75% of the planned dosage of lenvatinib during Cycle 1 as a result of treatment-related failure.
Time Frame: Cycle 1 (4 weeks) of each dose level
Population: ITT/ safety population included all participants who received at least one dose of lenvatinib.
Measure: Number; unit: Participants
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Participants
  Febrile neutropenia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Thrombocytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypertension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Secondary Outcome: Treatment-Related Adverse Events (All Grades) With an Overall Incidence Greater Than or Equal to 10%
Description: Treatment-related AEs were untoward medical events that were considered by the investigator to be possibly or probably related to lenvatinib.
Time Frame: First date of study treatment to date of withdrawal from study or last dose of study treatment, up to approximately 13 years and 8 months
Population: Safety population (ITT population) included all participants who took at least one dose of lenvatinib.
Measure: Number; unit: Percentage of participants
Groups:
- Lenvatinib 0.2 - 6.4 mg; Lenvatinib 12 - 20 mg: Lenvatinib tablets (at the appropriate dose for a given dose level) were taken orally, once daily on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided).
- Lenvatinib 25 mg: Two 10 mg lenvatinib tablets and five 1.0 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided).
- Lenvatinib 32 mg: Three 10 mg lenvatinib tablets and two 1.0 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided).
Arm/Group | Lenvatinib 0.2 - 6.4 mg | Lenvatinib 12 - 20 mg | Lenvatinib 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 21 | 30 | 24 | 7
Percentage of participants
  Hypertension | 10 | 40 | 63 | 57
  Nausea | 38 | 17 | 58 | 43
  Diarrhoea | 19 | 27 | 50 | 57
  Stomatitis | 5 | 20 | 63 | 57
  Proteinuria | 14 | 27 | 29 | 43
  Vomiting | 33 | 10 | 33 | 14
  Lethargy | 14 | 17 | 38 | 29
  Dysphonia | 0 | 13 | 46 | 43
  Dry skin | 5 | 10 | 46 | 14
  Fatigue | 10 | 23 | 21 | 14
  Anorexia | 10 | 17 | 21 | 29
  Constipation | 10 | 10 | 33 | 14
  Headache | 0 | 7 | 29 | 29
  Abdominal pain | 0 | 7 | 29 | 0

5. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was the best confirmed response of complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD), or not evaluable (NE), recorded from the start of lenvatinib until disease progression/recurrence or death. CR; disappearance of all target lesions for at least 1 month. PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD; a 20% or greater increase in the sum of the longest diameter of measured lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions. SD; PR failed to be achieved in the overall response assessment and there was no PD observed at 7 weeks or later after starting lenvatinib.
Time Frame: Baseline to first date of documented CR, PR, SD, or PD, assessed up to approximately 4 years
Population: ITT population included all participants who received at least one dose of lenvatinib.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Percentage of participants
  Partial response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 33.3 | 12.5 | 28.6
  Stable disease | 0 | 0 | 25.0 | 33.3 | 66.7 | 0 | 33.3 | 55.6 | 83.3 | 33.3 | 66.7 | 42.9
  Progressive disease | 50.0 | 50.0 | 0 | 0 | 0 | 33.3 | 41.7 | 11.1 | 16.7 | 0 | 8.3 | 0
  Not evaluable | 25.0 | 0 | 0 | 0 | 0 | 0 | 8.3 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Lenvatinib
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: Pharmacokinetic (PK) population included all participants in the ITT/Safety population that had evaluable PK data in at least one treatment cycle. The PK analysis set where data at specified timepoints was available.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 11 | 9 | 6 | 3 | 24 | 7
  Cycle 1 Day 1 | 0.753 (0.2176) | 1.740 (0.6921) | 4.255 (1.7474) | 20.967 (11.6741) | 49.883 (15.9952) | 127.067 (91.3320) | 259.990 (108.1789) | 209.004 (112.0090) | 375.077 (158.1811) | 408.797 (105.6923) | 630.589 (234.1659) | 649.927 (237.7462)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 2.385 (0.5162) | 5.477 (1.5988) | 9.610 (2.3193) | 36.483 (10.9339) | 92.137 (29.0365) | 197.217 (136.7307) | 291.414 (146.1972) | 187.467 (86.3962) | 368.937 (148.8160) | 238.670 (NA) — not evaluable, n=1 | 544.718 (183.1259) | 562.416 (121.4056)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Lenvatinib
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: PK population included all participants in the ITT/Safety population that had evaluable PK data in at least one treatment cycle. The PK analysis set where data at specified timepoints was available.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 4 | 4 | 3 | 3 | 3 | 11 | 9 | 6 | 3 | 24 | 7
  Cycle 1 Day 1 | 4.280 (1.440) | 5.785 (2.569) | 3.263 (1.194) | 3.973 (3.494) | 9.557 (12.658) | 2.023 (1.035) | 2.348 (1.144) | 1.897 (0.7768) | 2.287 (0.3881) | 2.533 (0.826) | 1.770 (0.715) | 2.674 (2.038)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 2 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 2.225 (0.3889) | 2.680 (0.589) | 13.475 (14.814) | 2.360 (1.179) | 2.173 (0.583) | 2.103 (0.405) | 2.021 (1.295) | 1.944 (0.604) | 2.352 (0.705) | 3.000 (NA) — not evaluable n=1 | 2.983 (1.481) | 1.500 (0.408)

8. Secondary Outcome: Apparent Plasma Half-life (t1/2) of Lenvatinib
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 11 | 9 | 6 | 3 | 24 | 7
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 2 | 3 | 10 | 9 | 6 | 3 | 23 | 6
  Cycle 1 Day 1 |  |  | 18.180 (11.342) | 10.695 (8.789) | 12.805 (3.118) | 8.077 (0.749) | 5.981 (0.4840) | 6.567 (0.9553) | 7.115 (1.0866) | 6.960 (1.230) | 5.848 (1.018) | 5.550 (0.599)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 29.540 (8.2731) | 26.380 (8.0427) | 20.840 (NA) — Not evaluable n=1 | 10.827 (5.555) | 9.973 (1.288) | 8.330 (0.517) | 6.935 (1.1681) | 6.829 (1.019) | 6.935 (0.9313) | 8.090 (NA) — Not evaluable n=1 | 6.025 (0.704) | 6.675 (0.5216)

9. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 to Infinity (AUC(0-inf))
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
nanogram*hour per milliliter (ng*hr/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 2 | 3 | 10 | 9 | 6 | 3 | 23 | 6
  Cycle 1 Day 1 |  |  | 123.745 (20.810) | 376.645 (312.1240) | 780.275 (189.116) | 1335.493 (894.562) | 1895.454 (467.145) | 1693.298 (1011.7941) | 3683.590 (2210.4521) | 4238.680 (2602.9271) | 4413.263 (1946.571) | 4383.678 (1697.248)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 99.325 (0.1202) | 174.310 (46.259) | 370.390 (NA) — Not evaluable n=1 | 585.247 (397.909) | 1150.393 (192.365) | 1952.430 (1323.783) | 2278.016 (851.258) | 1558.101 (760.687) | 3310.673 (1544.708) | 2260.040 (NA) — Not evaluable n=1 | 4549.825 (1161.045) | 4391.160 (997.486)

10. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 to 24 Hours (AUC(0-24))
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 11 | 9 | 6 | 3 | 24 | 7
  Cycle 1 Day 1 | 14.348 (4.500) | 30.207 (14.521) | 61.915 (17.164) | 220.910 (129.838) | 659.553 (209.129) | 1168.257 (799.169) | 1655.035 (555.479) | 1537.476 (876.6805) | 3250.843 (1826.8789) | 3709.550 (2059.6379) | 4074.803 (1666.2780) | 4601.014 (1887.3642)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 43.305 (8.5913) | 85.477 (37.054) | 199.100 (NA) — Not evaluable n=1 | 422.873 (270.528) | 931.307 (179.514) | 1691.160 (1167.750) | 2052.965 (789.504) | 1422.584 (697.699) | 2947.920 (1286.805) | 1934.500 (NA) — Not evaluable n=1 | 4224.095 (1120.837) | 4020.185 (899.182)

11. Secondary Outcome: Clearance Corrected for the Fraction of Lenvatinib Absorbed (CL/F)
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liter per hour (L/hr)
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Liter per hour (L/hr)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 2 | 3 | 10 | 9 | 6 | 3 | 23 | 6
  Cycle 1 Day 1 |  |  | 6.560 (1.103) | 6.470 (5.360) | 4.225 (1.0253) | 8.190 (7.923) | 6.614 (1.336) | 9.534 (4.307) | 6.157 (4.240) | 5.980 (3.236) | 6.863 (3.354) | 8.827 (5.058)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 4.710 (0.9334) | 5.200 (1.802) | 4.020 (NA) — Not evaluable n=1 | 5.347 (3.942) | 3.533 (0.747) | 5.557 (4.200) | 6.896 (3.360) | 10.110 (3.321) | 6.437 (3.668) | 10.340 (NA) — Not evaluable n=1 | 6.378 (2.302) | 7.978 (2.763)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Liter (L)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 2 | 3 | 10 | 9 | 6 | 3 | 23 | 6
  Cycle 1 Day 1 |  |  | 162.975 (78.383) | 65.795 (0.6435) | 80.365 (37.922) | 97.190 (95.442) | 57.039 (11.887) | 88.069 (38.174) | 58.408 (32.346) | 56.350 (22.932) | 55.263 (22.411) | 68.073 (32.456)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 1 | 3 | 3 | 3 | 8 | 7 | 6 | 1 | 4 | 4
  Cycle 2 Day 1 | 206.360 (96.068) | 208.937 (114.969) | 120.810 (NA) — Not evaluable n=1 | 65.437 (24.894) | 51.487 (16.805) | 67.747 (51.897) | 70.881 (40.419) | 99.960 (37.787) | 60.683 (26.763) | 120.730 (NA) — Not evaluable n=1 | 57.143 (28.550) | 76.610 (25.967)

13. Secondary Outcome: Fraction of Unchanged Lenvatinib Excreted in the Urine (fe)
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of lenvatinib
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
Percentage of lenvatinib
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 4 | 3 | 3 | 2 | 2 | 10 | 8 | 6 | 3 | 20 | 7
  Cycle 1 Day 1 | 0.530 (0.0141) | 0.253 (0.0457) | 0.217 (0.0896) | 0.363 (0.1290) | 0.355 (0.0354) | 0.390 (0.0849) | 0.487 (0.3137) | 0.783 (0.7928) | 0.348 (0.1910) | 0.690 (0.4851) | 0.576 (0.3042) | 0.503 (0.3004)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 2 | 2 | 1 | 3 | 7 | 6 | 4 | 1 | 5 | 3
  Cycle 2 Day 1 | 1.240 (NA) — Not evaluable n=1 | 0.715 (0.1626) | 0.605 (0.0636) | 0.535 (0.3748) | 1.050 (NA) — Not evaluable n=1 | 0.557 (0.2212) | 0.689 (0.4208) | 0.663 (0.2873) | 0.825 (0.2786) | 0.630 (NA) — Not evaluable n=1 | 0.778 (0.3801) | 0.527 (0.1595)

14. Secondary Outcome: Renal Clearance (CLr) of Lenvatinib
Time Frame: Cycles 1 and 2 Day 1: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 3 | 3 | 12 | 9 | 6 | 3 | 24 | 7
L/hour
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 2 | 10 | 8 | 6 | 3 | 20 | 7
  Cycle 1 Day 1 | 0.060 (0.0064) | 0.037 (0.0167) | 0.027 (0.0042) | 0.035 (0.0233) | 0.021 (0.0113) | 0.017 (0.0078) | 0.039 (0.0243) | 0.064 (0.0534) | 0.020 (0.0095) | 0.046 (0.0466) | 0.041 (0.0233) | 0.035 (0.0144)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 1 | 2 | 1 | 3 | 7 | 6 | 4 | 1 | 4 | 3
  Cycle 2 Day 1 | 0.050 (NA) — Not evaluable n=1 | 0.045 (0.011) | 0.022 (NA) — Not evaluable n=1 | 0.029 (0.0042) | 0.034 (NA) — Not evaluable n=1 | 0.025 (0.0097) | 0.050 (0.0304) | 0.069 (0.021) | 0.048 (0.36) | 0.065 (NA) — Not evaluable n=1 | 0.52 (0.019) | 0.045 (0.0247)

15. Secondary Outcome: Effect of Food on the Area Under the Curve From Zero to 24 Hours (AUC(0-24))
Time Frame: Cycle 1 Day 15 and Day 22: 0-24 hours postdose (Cycle length = 28 days)
Population: The Food Effect Population consisted of all participants who agreed to participate in this part of the study, have received both the Day 15 and Day 22 doses, with PK sampling during 24 hours following those doses and consumed at least half (approximately) of the high fat breakfast when in the fed period.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Lenvatinib Fed 25 mg; Lenvatinib Fasted 25 mg: Participants who agreed to participate in the food-effect study received a single oral dose of lenvatinib (25 mg) after a high-fat meal (including potatoes and bacon) or following at least a 10 hour fast on the morning of either Cycle 1 Day 15 or Cycle 1 Day 22 between 8:00 am and 10:00 am. Whichever state (fed or fasted) the participant took the lenvatinib on Day 15, they did the opposite on Day 22. All other doses were taken on an empty stomach after waking, followed by fasting for 2 hours with only clear liquids allowed.
Arm/Group | Lenvatinib Fed 25 mg | Lenvatinib Fasted 25 mg
Number analyzed (Participants) | 11 | 11
ng*hr/mL | 3851.773 (993.1449) | 4039.681 (1567.4169)

16. Secondary Outcome: Effect of Food on the Maximum Plasma Concentration (Cmax) of Lenvatinib
Time Frame: Cycle 1 Day 15 and Day 22: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib Fed 25 mg | Lenvatinib Fasted 25 mg
Number analyzed (Participants) | 11 | 11
ng/mL | 508.558 (165.7591) | 544.058 (248.5409)

17. Secondary Outcome: Effect of Food on Time to Maximum Concentration (Tmax) of Lenvatinib
Time Frame: Cycle 1 Day 15 and Day 22: 0-24 hours postdose (Cycle length = 28 days)
Population: as for outcome 15
Measure: Median (Full Range); unit: Hours
Groups:
- Lenvatinib Fed State 25 mg; Lenvatinib Fasted State 25 mg: Participants who agreed to participate in the food-effect study received a single oral dose of lenvatinib (25 mg) after a high-fat meal (including potatoes and bacon) or following at least a 10 hour fast on the morning of either Cycle 1 Day 15 or Cycle 1 Day 22 between 8:00 am and 10:00 am. Whichever state (fed or fasted) the participant took the lenvatinib on Day 15, they did the opposite on Day 22. All other doses were taken on an empty stomach after waking, followed by fasting for 2 hours with only clear liquids allowed.
Arm/Group | Lenvatinib Fed State 25 mg | Lenvatinib Fasted State 25 mg
Number analyzed (Participants) | 11 | 11
Hours | 4.980 [2.00 to 5.07] | 2.030 [1.00 to 3.07]
Statistical Analysis 1: Comparison: Lenvatinib Fed State 25 mg vs Lenvatinib Fasted State 25 mg; This was a pilot study and a statistical sample size calculation was not performed; Test type: Superiority or Other; p = 0.0146, Wilcoxon signed-rank test

18. Other Pre Specified Outcome: Pharmacodynamic (PD) Biomarkers of Lenvatinib in Peripheral Blood Mononuclear Cells (PBMCs) and Tumor Samples
Description: Based on the data in assay development stage before PD biomarker analysis in study E7080-E044-101 we did not find the appropriate PD biomarker in PBMC, therefore we did not have any biomarker analysis for PK/PD analysis.
Time Frame: Blood: Cycle 1 Day 1, Day 15, or Day 22, Cycle 2 Day 1 Tumor tissue: Screening and after at least one 28-day Cycle of study treatment
Population: No appropriate PD biomarker in PBMC, therefore we did not have any biomarker analysis for PK/PD analysis.
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib Fasted/Fed 25 mg | Lenvatinib Fed/Fasted 25 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected for up to approximately 13 years and 8 months
Description: Treatment-emergent adverse events were defined as AEs that emerged during treatment, having been absent at pre-treatment, or that worsened in severity relative to the pre-treatment state, or occurred within 30 days of last dose of the treatment. Only treatment-emergent AEs and SAEs were reported.
Groups:
- Lenvatinib 6.4 mg: Six 1.0 mg lenvatinib tablets and four 0.1 mg lenvatinib tablets were taken orally, once daily. Lenvatinib was to be taken on an empty stomach shortly after waking. Participants were fasted for 2 hours following administration of lenvatinib and could drink only clear fluids during this time (grapefruit juice was to be avoided). If 1 of 3 participants experienced DLT during Cycle 1 (4 weeks) an additional 3 participants were to be treated at this dose level. If 5 of the 6 participants in the expanded dose level did not experience DLT during the first 4 weeks of therapy, no additional DLT was observed, the next dose level was opened for enrollment. If more than 1 participant experienced DLT during the first 4 weeks of therapy, dose escalation was stopped and theMTD was determined. An additional 12 participants were treated at the MTD level.
Arm/Group | Lenvatinib 0.2 mg | Lenvatinib 0.4 mg | Lenvatinib 0.8 mg | Lenvatinib 1.6 mg | Lenvatinib 3.2 mg | Lenvatinib 6.4 mg | Lenvatinib 12 mg | Lenvatinib 12.5 mg | Lenvatinib 16 mg | Lenvatinib 20 mg | Lenvatinib Fasted/Fed 25 mg | Lenvatinib Fed/Fasted 25 mg | Lenvatinib (MTD Cohort) 25 mg | Lenvatinib 32 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/4 | 1/4 | 1/3 | 0/3 | 2/3 | 1/12 | 1/9 | 1/6 | 3/3 | 0/6 | 0/5 | 3/24 | 2/7
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 1/4 | 1/3 | 0/3 | 3/3 | 5/12 | 4/9 | 2/6 | 3/3 | 2/6 | 2/5 | 15/24 | 3/7
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 3/3 | 3/3 | 3/3 | 12/12 | 9/9 | 6/6 | 3/3 | 6/6 | 5/5 | 24/24 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 0.2 mg (N=4) | Lenvatinib 0.4 mg (N=4) | Lenvatinib 0.8 mg (N=4) | Lenvatinib 1.6 mg (N=3) | Lenvatinib 3.2 mg (N=3) | Lenvatinib 6.4 mg (N=3) | Lenvatinib 12 mg (N=12) | Lenvatinib 12.5 mg (N=9) | Lenvatinib 16 mg (N=6) | Lenvatinib 20 mg (N=3) | Lenvatinib Fasted/Fed 25 mg (N=6) | Lenvatinib Fed/Fasted 25 mg (N=5) | Lenvatinib (MTD Cohort) 25 mg (N=24) | Lenvatinib 32 mg (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib 0.2 mg (N=4) | Lenvatinib 0.4 mg (N=4) | Lenvatinib 0.8 mg (N=4) | Lenvatinib 1.6 mg (N=3) | Lenvatinib 3.2 mg (N=3) | Lenvatinib 6.4 mg (N=3) | Lenvatinib 12 mg (N=12) | Lenvatinib 12.5 mg (N=9) | Lenvatinib 16 mg (N=6) | Lenvatinib 20 mg (N=3) | Lenvatinib Fasted/Fed 25 mg (N=6) | Lenvatinib Fed/Fasted 25 mg (N=5) | Lenvatinib (MTD Cohort) 25 mg (N=24) | Lenvatinib 32 mg (N=7)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (3) | 3 (7) | 2 (2) | 3 (9) | 2 (2) | 2 (3) | 3 (3) | 4 (4) | 5 (9) | 17 (29) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 3 (4) | 3 (8) | 3 (3) | 3 (6) | 5 (9) | 4 (12) | 16 (36) | 4 (12)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 3 (4) | 1 (1) | 5 (5) | 3 (5) | 15 (23) | 4 (8)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (3) | 1 (1) | 3 (7) | 0 (0) | 4 (7) | 4 (6) | 1 (2) | 2 (2) | 1 (1) | 4 (9) | 13 (28) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (8) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 13 (20) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 10 (17) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (2) | 4 (7) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 5 (8) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (6) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (8) | 1 (1) | 3 (5) | 3 (4) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 10 (21) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 9 (18) | 4 (7)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 3 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 3 (7) | 3 (9) | 2 (4) | 1 (1) | 4 (7) | 2 (4) | 8 (13) | 3 (5)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 3 (3) | 7 (9) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (5) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 10 (14) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 2 (4) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 7 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (12) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 3 (3) | 12 (14) | 3 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 7 (9) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 5 (9) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (6) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 11 (15) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 5 (7) | 2 (4) | 4 (11) | 1 (2) | 4 (6) | 2 (4) | 15 (24) | 4 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 4 (4) | 1 (3) | 2 (2) | 1 (2) | 3 (4) | 12 (19) | 3 (4)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 3 (8) | 2 (6) | 1 (3) | 0 (0) | 7 (22) | 3 (19)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (4) | 2 (10) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 2 (5) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound closure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No